CLINICAL TRIAL: NCT05982977
Title: Study on the Effect Mechanism of Acupuncture Combined With Swallowing Training to Regulate the Cortical Swallowing Network in Oral Dysphagia of Stroke
Brief Title: Study on the Effect Mechanism of Acupuncture Combined With Swallowing Training in Oral Dysphagia of Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qingqing Zhang (Other)
Collaborators: Fujian University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Qingqing Zhang, Lecturer, Fujian University of Traditional Chinese Medicine
Organization: Fujian University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022J01880
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Dysphagia; Stroke; Oral Phase
Keywords: Dysphagia; stroke; cortical swallowing network; Oral Phase
MeSH Terms: conditions — Deglutition Disorders; Stroke | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: This study was a parallel, randomized controlled trial. Qualified subjects were numbered according to the inclusion order and randomly assigned to the swallowing training treatment group and the acupuncture combined swallowing training treatment group in a 1:1 ratio.
Who Masked: Outcomes Assessor
Masking Description: Since acupuncture intervention could not blind subjects and investigators, evaluators and statisticians were secretly grouped to avoid measurement bias as much as possible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture rehabilitation group (Experimental): Acupuncture rehabilitation intervention was given on the basis of conventional rehabilitation therapy.Disinfected with 75% alcohol and applied the needles at a depth of 25-35mm. Acupuncture stimulation of Lianquan (CV23) and Fengchi (GB20). The needles were retained for 30 minutes/time, once a day, and 5 days/week for a total of 4 weeks.
  Interventions: Other: Acupuncture
- Conventional rehabilitation group (Active Comparator): This group participants would take swallowing training 30 minutes/time, once a day, 5 days/week, a total of 4 weeks of intervention. At the same time, stroke basic treatment, nutritional support and other symptomatic treatment
  Interventions: Behavioral: Conventional rehabilitation

INTERVENTIONS:
Other: Acupuncture — The patient was placed in a supine position, selected Lianquan, Fengchi, and acupoints.
  Arms: Acupuncture rehabilitation group
Behavioral: Conventional rehabilitation — swallowing training included breathing training, masticatory muscle training, oral movement training and feeding training.
  Arms: Conventional rehabilitation group

SUMMARY:
Up to 84% of patients after stroke are accompanied by dysphagia, of which 53% are oral dysphagia. The oral phase is the initial phase of swallowing activity and the only stage of swallowing that is completely discretionary. Swallowing activity in the oral stage is not only related to the formation and push of food pellets, but also affects the continuity between the transition from spontaneous swallowing to the swallowing reflex.

DETAILED DESCRIPTION:
After stroke, patients are prone to oral dysphagia, poor control of food masses and liquids in the mouth, resulting in food spillover, residual and premature overflow, resulting in dehydration, malnutrition, aspiration, pneumonia and other serious consequences, which greatly reduce the eating safety and quality of life of patients after stroke. Therefore, the rehabilitation of oral swallowing function is a way for patients with swallowing disorder after stroke to return to society and improve their quality of life. Previous studies have found that acupuncture is an effective intervention to improve swallowing disorder in oral stage after stroke. Whether acupuncture promotes the improvement of swallowing function in oral stage by regulating the synergic activity of cortical swallowing network and muscle group has not been fully clarified.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting the diagnostic criteria for acute ischemic stroke established by the Neurology Society of the Chinese Medical Association and confirmed by craniocerebral CT or MRI;
2. Oral dysphagia caused by stroke;
3. Currently diet is restricted, FOIS score is 5 or less; WST score 3 or above;
4. MoCA score of 21 or above, able to understand and follow simple instructions from the treatment staff, able to cooperate and willing to undergo examination and treatment;
5. 40 to 75 years old;
6. Conscious and stable vital signs;
7. Convalescent patients with stroke course and dysphagia duration between 1-6 months;
8. Voluntary participation and informed consent.

Exclusion Criteria:

1. Patients with dysphagia not caused by stroke or non-stroke oral dysphagia;
2. Previous history of stroke or dysphagia;
3. Patients with serious primary diseases or mental disorders of other systems;
4. Suffering from various bleeding prone diseases;
5. Severe needle fainting;
6. People with metal implants.
7. Patients with poor compliance are not treated as prescribed

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Oral functional score | 4 weeks (Before and after intervation)
  To assess participants' oral swallowing function

SECONDARY OUTCOMES:
Surface electromyography | 4 weeks (Before and after intervation)
  To assess the swallowing muscle activity
Water swallowing test (WST) | 4 weeks (Before and after intervation)
  The severity of dysphagia was assessed by the WST. Level 1: Can drink 30ml water successfully within 5 seconds; Level 2: Drink water more than 2 times, can swallow without choking. Level 3: Can be drunk once, but cough. Level 4: swallowed more than twice, but with choking. Level 5: Frequent choking, unable to swallow all. Normal: Level 1, Suspicious: Level 1, more than 5 seconds or level 2; Abnormal: Level 3 to 5
Standardized Swallowing Assessment (SSA) | 4 weeks (Before and after intervation)
  To assess the severity of swallowing. The lowest score on this scale is 18 points, the highest score is 46 points, the higher the score, the worse the swallowing function.
Functional Oral Intake Scale (FOIS) | 4 weeks (Before and after intervation)
  To assess the condition of swallowing. The grade of FOIS was categorized as level 1 to 3 (poor FOIS: tube feeding), levels 4 and 5 (moderate FOIS: total oral diet requiring special preparation) or levels 6 and 7 (good FOIS: total oral diet without special preparation).
Teacher salivation rating (TDS) | 4 weeks (Before and after intervation)
  Assess salivation. Level 1: No salivation; Level 2: Small amount, occasional flow. Level 3: Stream from time to time; Level 4: Flow frequently, but not linearly; Level 5: Flow in line, chest often wet
Swallowing Related Daily Quality of Life Scale (SWAL-QOL) | 4 weeks (Before and after intervation)
  Assessed patients' quality of life. The SWAL-QOL scale consists of 11 dimensions, covering 44 items, of which 10 dimensions measure patients' quality of life and one dimension measures patients' swallowing symptoms. The 10 quality of life dimensions included 30 items, of which 8 (25 items in total) were related to swallowing, including psychological burden, eating time, appetite, food choice, verbal communication, fear of eating, mental health, and social interaction: the common dimension had 2 (5 items in total), including fatigue and sleep. The dimension of swallowing symptoms included 14 items. The SWAL-OOL scale was scored by Likert scoring method. The higher the score of five levels (1-5 respectively), the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Zhang, Principal Investigator — Fujian University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No